CLINICAL TRIAL: NCT00002735
Title: Induction Chemotherapy Followed By Chemoradiation For Organ Preservation In Patients With Advanced Resectable Cancer Of The Hypopharynx And Base Of Tongue, Phase II
Brief Title: SWOG-9451, Combination Chemo & RT For Patients With Stage III/Stage IV Cancer of the Hypopharynx or Tongue
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to poor accrual.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000064634; SWOG-9451 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-09-01 (Estimated); Last update posted 2015-09-30 (Estimated); Status verified 2015-09

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Induction Chemotherapy; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): induction chemotherapy followed by chemoradiation
  Interventions: Drug: Induction chemotherapy; Drug: cisplatin; Drug: fluorouracil; Radiation: low-LET cobalt-60 gamma ray therapy

INTERVENTIONS:
Drug: Induction chemotherapy — Cisplatin and 5-Fluorouracil
  Other Names: platinol; 5-FU
Drug: cisplatin — Cisplatin 100 mg/m2 IV infusion over 90 minutes Day 1 every 21 days for 2 cycles.
  Other Names: platinol
Drug: fluorouracil — 5-Fluorouracil 1,000 mg/m2/day continuous IV infusion over 24 hours Days 1 through 5 every 21 days for 2 cycles.
  Other Names: 5-FU
Radiation: low-LET cobalt-60 gamma ray therapy — 180 cGy per day, Days 1-5, every week for eight weeks
  Other Names: RT

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and radiation therapy in treating patients with stage III or stage IV cancer of the hypopharynx or tongue.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete histologic response rate (which represents the rate of organ preservation) to induction with cisplatin/fluorouracil followed by radiotherapy plus cisplatin in patients with selected stage III/IV cancer of the hypopharynx or base of the tongue. II. Evaluate the feasibility of accruing and treating patients with this regimen in a multi-institutional setting. III. Determine the overall complete response rate in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to center and tumor site (hypopharynx vs base of tongue). Base of tongue stratum closed as of November 15, 1998. Regimen A: Patients receive cisplatin IV over 90 minutes on days 1 and 22 and fluorouracil IV over 120 minutes on days 1-5 and 22-26. Patients with measurable neck nodes discontinue therapy if disease has progressed by day 22. All patients who achieve complete or partial response at day 43 proceed to regimen B. All others proceed to resection followed by radiotherapy (off study). Regimen B (begins within 3-4 weeks of start of second induction course): Patients receive cisplatin IV over 90 minutes every 3 weeks for 3 courses. Concurrently, patients receive radiotherapy 5 days a week for 5.6 weeks. Patients are reassessed at 8-12 weeks after radiotherapy. Patients who are disease free are observed. Other patients undergo surgical resection of nodes and/or primary tumor. Patients are followed every 4-6 weeks for 1 year, every 2 months for 1 year, every 4 months for 2 years, every 6 months for 1 year, then annually thereafter.

PROJECTED ACCRUAL: Up to 70 patients (35/tumor site) will be accrued for this study over 3.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed squamous cell carcinoma of the hypopharynx or base of the tongue that is newly diagnosed and considered resectable For hypopharyngeal cancer, total laryngectomy would be required surgery Disease staged by clinical exam, endoscopy, and CT or MRI Stage III that is T2-3 N0-1 M0 Stage IV that is T2-3 N2-3 M0 Measurable or evaluable disease other than pleural effusion, ascites, or disease documented by indirect evidence Closed to patients with cancer of the base of tongue as of 11/15/1998

PATIENT CHARACTERISTICS: Age: Adult Performance status: SWOG 0 or 1 Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 times normal AST or ALT no greater than 3 times normal Renal: Creatinine no greater than 2 times normal Creatinine clearance at least 60 mL/min Magnesium normal (supplementation allowed) Other: Average hearing loss in both ears no greater than 40 dB in 50-2,000 Hz range No second malignancy within 5 years except: Adequately treated nonmelanomatous skin cancer Carcinoma in situ of the cervix Stage I/II cancer (other than head/neck) in complete remission Not pregnant or nursing Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: No prior therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 1996-04; Primary Completion 2004-04 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Complete response | 23 to 27 weeks after beginning treatment
  Complete disappearance of all measurable and evaluable disease. No new lesions, No disease related symptoms. No evidence of non-evaluable disease, including normalization of markers and other abnormal lab values. Specifically, the rate of organ preservation (no surgery required at the primary tumor site).

CONTACTS AND LOCATIONS:
Overall Officials: Susan G. Urba, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (18):
- United States (18):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Colorado Cancer Center, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - Veterans Affairs Medical Center - Brooklyn, Brooklyn, New York
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - University of Texas Medical Branch, Galveston, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas

REFERENCES:
- [Result] Urba SG, Moon J, Giri PG, Adelstein DJ, Hanna E, Yoo GH, Leblanc M, Ensley JF, Schuller DE. Organ preservation for advanced resectable cancer of the base of tongue and hypopharynx: a Southwest Oncology Group Trial. J Clin Oncol. 2005 Jan 1;23(1):88-95. doi: 10.1200/JCO.2005.04.017. PMID 15625363
- [Result] Urba S, Moon J, LeBlanc M, et al.: Induction chemotherapy followed by chemoradiation for organ preservation in patients (pts) with advanced resectable cancer of the base of tongue (BOT) and hypopharynx (HP): a Southwest Oncology Group trial. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-919, 2002.